CLINICAL TRIAL: NCT02749097
Title: A PHASE I, RANDOMIZED, PLACEBO-CONTROLLED, SINGLE DOSE ESCALATION STUDY TO INVESTIGATE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF SHR0534 IN HEALTHY VOLUNTEERS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0534A001
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
MeSH Terms: interventions — SHR0534

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Cohort 1 (Experimental): Single oral dose of 10 mg SHR0534 or matching placebo
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 2 (Experimental): Single oral dose of 25 mg SHR0534 or matching placebo
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 3 (Experimental): Single oral dose of 50 mg SHR0534 or matching placebo
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 4 (Experimental): Single oral dose of 100 mg SHR0534 or matching placebo
  Interventions: Drug: SHR0534; Drug: Placebo
- Cohort 5 (Experimental): Single oral dose of 200 mg SHR0534 or matching placebo
  Interventions: Drug: SHR0534; Drug: Placebo

INTERVENTIONS:
Drug: SHR0534
Drug: Placebo

SUMMARY:
This is a randomized, placebo-controlled, single dose escalation study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR0534. The study will be conducted with starting dose of 10 mg followed by dose escalation groups up to 200 mg. Eight subjects will be randomized in 3:1 ratio in each cohort to receive the study drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be adequately informed of the nature and risks of the study, able to understand the risks associated with the study, and are willing to provide written informed consent prior to screening.
* Must have be at least 50 kg (110 lb), and a BMI between 19.0 to 32.0 kg/m2, inclusive.
* Drug screen (including alcohol) must have been negative at Screening and on admission to study site.
* Subjects must be free of any clinically significant diseases based on medical history , physical examination and/or the investigator's judgment
* Clinical laboratory tests (i.e. CBC, platelet count, blood chemistries, and urinalysis) must be within the normal reference range or clinically acceptable as determined by the investigator.
* Completion of the screening process within 14 days prior to dosing.
* Must be able to communicate effectively with the study personnel.
* Must be nonsmokers, defined as not having smoked tobacco or used chewing tobacco or nicotine-containing products in the 6 months prior to Day 1. Cotinine test must be negative at Screening and Day -1.
* Must have, in the investigator's opinion, no clinically significant diseases or abnormal laboratory test values as determined by medical and psychiatric history, physical examination, or laboratory evaluations conducted at the screening visit or on clinic admission.
* Subjects of reproductive potential with partners who are women of childbearing potential, will be instructed to, and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 90 days after discontinuing treatment with the investigational product. Highly effective methods of birth control include sexual abstinence, vasectomy or a condom with spermicide (men) in combination with barrier methods, oral, injected, or implanted hormonal birth control methods, or placement of an intrauterine device or intrauterine system (for female partner).
* Subjects must agree not to donate sperm during the study and for 90 days after discontinuing treatment with the investigational product.

Exclusion Criteria:

* History of hypersensitivity to SHR0534 or its components.
* History of or current clinically important systemic illnesses, including but not limited to cardiovascular, pulmonary, hepatobiliary, renal, hematological, gastrointestinal, endocrinological, immunological, dermatological, neurological, or psychiatric diseases, or any conditions that may place the subject at increased risk as determined by the investigator.
* Any condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of surgery or major trauma within 12 weeks of study entry, or surgery planned during the study.
* History of allergy or hypersensitivity to heparin, or heparin-induced thrombocytopenia.
* History of myocardial infarction, stroke or sudden unexplained death in a first degree family member under the age of 60 years.
* History of liver disease. Those with ALT or AST >1.5 times upper limit of normal must be excluded.
* Subjects with anemia or abnormal hematology parameters with clinically significance as determined by the investigator must be excluded.
* History or presence of clinically significant electrocardiogram (ECG) abnormalities.
* History of alcohol dependent, habitual heavy users of caffeinated beverages judged by the investigator.
* Have used any alcohol-containing products within 3 days of Day 1.
* Urine drug screen test positive for ethanol, cocaine, tetrahydrocannabinol (THC), barbiturates, amphetamines, benzodiazepines, or opiates.
* Have used any drugs or substances (including herbal supplements) known to inhibit or induce cytochrome (CYP) P450 enzymes including CYP3A4, CYP2C8 and CYP2C9 within 28 days prior to the first dose and throughout the study.
* Use of any over-the-counter (OTC), nutraceuticals, or prescription medications (except as specified within this protocol) within 7 days or 5 half lives (whichever is longer), prior to receiving investigational product. By exception, up to 2 g per day acetaminophen (paracetamol) for analgesia will be allowed up to 48 hours prior to Day -1.
* Use of xanthine-containing substances, or alcohol-containing products within 48 hours prior to study drug administration.
* Use of grapefruit or related citrus fruit products 7 days prior to the study drug administration or intend to use during the study.
* Have taken other investigational drugs or participated in any clinical trial within 30 days prior to first dose of study drug in this study.
* Have had significant blood loss (>450 mL) or have donated 1 or more units of blood or plasma within 12 weeks prior to study entry.
* Have a positive test at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb).
* Have any other condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures.
* Any individual involved in the planning or conduct of this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From baseline up to 8 days after single dose

SECONDARY OUTCOMES:
Area under the plasma concentration curve (AUC) | From time 0 to 168 hours after single dose
Peak plasma concentration (Cmax) after dose after dose | From time 0 to 168 hours after single dose
Terminal elimination halflife (t½) for SHR0534 after single dose after dose | From time 0 to 168 hours after single dose
Changes in the concentrations of blood glucose after SHR0534 is orally administered | From baseline up to 8 hours after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ruff, M.D, Principal Investigator — ICON Development Solutions